CLINICAL TRIAL: NCT03403959
Title: The Neurobiology of Seasonal Affective Disorder: Exploring the High Prevalence in Severe Visual Impairment
Brief Title: Seasonal Affective Disorder and Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Helle Østergaard Madsen, MD, Psychiatric Centre Rigshospitalet
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BlindSAD
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Seasonal Affective Disorder; Visual Impairment
Keywords: pupillometry; light therapy; visual impairment; melatonin; ipRGC
MeSH Terms: conditions — Seasonal Affective Disorder; Vision Disorders | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: The study combines two models: a case/control study with observational outcomes where all cases are consequently included in a non-randomized interventional study
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor and the participant is unaware of ipRGC function prior to and during treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD (Experimental): Persons with visual impairment and SAD are assessed by clinical interview, depression rating, diurnal saliva melatonin and cortisol and chromatic pupillometry during symptomatic winter phase and asymptomatic summer phase. Winter assessment is followed by a 6 week light therapy protocol ending with assessment of depression severity and repeated pupillometry.
  Interventions: Device: light therapy
- non-SAD (No Intervention): Control participants with similar visual impairment but without SAD/sSAD are assessed by clinical interview, depression rating, diurnal saliva melatonin and cortisol and chromatic pupillometry in winter and summer.

INTERVENTIONS:
Device: light therapy — 6 weeks morning treatment with bright light therapy in own home.
  Arms: SAD

SUMMARY:
As a subtype of major depressive disorder, seasonal affective disorder (SAD) or winter depression causes severe reductions in both quality of life and productivity and results in high morbidity and frequent sick leave (1). SAD is a prevalent disorder with rates as high as 3-5% in central European countries and 8-10% in Scandinavian countries. In our recent screening survey among persons with severe visual impairment or blindness (visual acuity < 6/60), we found a strikingly high prevalence of SAD of 17 % compared to 8% in the fully sighted control group. Persons with maintained light perception had a highly increased SAD prevalence of 18 % whereas no light perception (NLP) respondents had an SAD prevalence of 13 %. Light is unquestionably of great importance in the development and treatment of SAD. It is suggested that a reduced retinal sensitivity to light leads to sub-threshold light input to the brain and consequently to the development of SAD. The novel retinal non-visual photoreceptors, the intrinsically photosensitive retinal ganglion cells (ipRGCs), are involved in the regulation of circadian rhythm and mood and their function are in part independent of the function of the classical rod and cone photoreceptors which form the basis of conscious visual perception. Function of the ipRGCs can be assessed by chromatic pupillometry where the sustained pupillary contractions following blue light stimulation (PIPR) is the main outcome. In persons with SAD without eye disorder the function of the ipRGCs is reduced. We here wish to investigate associations between ipRGC function and SAD symptoms, circadian profile and treatment response to light therapy in persons with visual impairment.

Persons with visual impairment (SAD and non-SAD) are assessed for ipRGC function with chromatic pupillometry, for seasonal mood variation by interview and questionnaire and for diurnal melatonin secretion by saliva analysis summer and winter. In winter SAD participants are treated with daily morning bright light for 6 weeks. Reduction in depression scores and tolerability is recorded.

ELIGIBILITY:
Inclusion Criteria:

Seasonal affective disorder. Visual impairment (Snellen visual acuity < 6/18) or visual field reduction (MD<10).

Exclusion Criteria:

Alcohol or drug abuse. Current or planned pregnancy. Other neuropsychiatric disorder. Antidepressant medication. Regular use of melatonin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
treatment response | 6 weeks
  Reduction in depression severity on the Structured interview guide for the Hamilton Depression Rating Scale - Seasonal affective disorder version (25 items version total score with range 0-78. Results from Hamilton Rating Scale for Depression 17 items (range 0-52) and the 8 item atypical symptom subscale (range 0-26) are reported. Higher scores indicate higher severity.
saliva melatonin concentration | 6 months
  Differences in melatonin secretion as indicated by area under curve (AUC) between SAD and non-SAD (summer and winter).

SECONDARY OUTCOMES:
PIPR - light therapy | 6 weeks
  Correlation between treatment response and ipRGC function as measured by the sustained (10-20 seconds) post-illumination pupillary contraction following blue light stimulation

OTHER OUTCOMES:
feasibility of light therapy | 6 weeks
  side effects and tolerability of light therapy
Late sustained post-illumination pupillary response to blue light | 6 months
  Difference in late PIPR (10-30 seconds post-illumination) following high intensity blue light between SAD and non-SAD and between seasons

CONTACTS AND LOCATIONS:
Overall Officials: Helle Ø Madsen, MD, Principal Investigator — Mental Health Center Copenhagen
Locations (1):
- Mental Health Center Copenhagen, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No